CLINICAL TRIAL: NCT02510547
Title: Comparison of a CrossBoss First Versus Standard Wire Escalation Strategy for Crossing Coronary Chronic Total Occlusion: the "CrossBoss First" Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Collaborators: Henry Ford Hospital (Other); Massachusetts General Hospital (Other); North Central Heart-Avera Sacred Heart Hospital (Unknown); Saint Lukes Hospital Mid America Heart Institute (Unknown); Missouri Heart Center (Unknown); University of Washington (Other); Deborah Heart and Lung Center (Other); Minneapolis Heart Institute (Other); Wellspan Heart and Vascular (Unknown); United Heart and Vascular Clinic and United Hospital (Unknown)
Responsible Party: Principal Investigator, Emmanouil Brilakis, Emmanouil Brilakis, MD, PhD, North Texas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-010
Record Dates: First submitted 2015-07-22; First posted 2015-07-29 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Arteriosclerosis; Coronary Artery Disease; Myocardial Ischemia; Coronary Disease
MeSH Terms: conditions — Arteriosclerosis; Coronary Artery Disease; Myocardial Ischemia; Coronary Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CrossBoss Catheter (Active Comparator): Crossing the CTO with upfront use of the CrossBoss catheter
  Interventions: Procedure: CrossBoss Catheter
- Antegrade Wire Escalation Strategy (Active Comparator): Crossing the CTO with upfront antegrade wire escalation strategy
  Interventions: Procedure: Antegrade Wire Escalation Strategy

INTERVENTIONS:
Procedure: CrossBoss Catheter — Upfront use of the CrossBoss catheter for CTO lesion crossing
  Arms: CrossBoss Catheter
Procedure: Antegrade Wire Escalation Strategy — Upfront guidewire escalation strategy for CTO lesion crossing
  Arms: Antegrade Wire Escalation Strategy

SUMMARY:
CrossBoss First is a single-blind randomized controlled trial that will randomize 246 patients undergoing clinically-indicated Chronic Total Occlusion Percutaneous Coronary Intervention, to upfront use of the CrossBoss catheter vs. antegrade guidewire escalation strategy The "CrossBoss First" study has two primary objectives. The primary efficacy objective is to compare the procedure time required to cross the CTO or abort the procedure with a CrossBoss first vs. antegrade wire escalation strategy. The investigators hypothesize that upfront use of the CrossBoss catheter will be associated with shorter procedure time required for CTO crossing compared with an antegrade wire escalation strategy.

The primary safety objective is to compare the frequency of procedural major adverse cardiovascular events (MACE) with upfront use of CrossBoss vs. a guidewire escalation strategy. The investigators hypothesize that upfront use of the CrossBoss catheter will be associated with similar incidence of MACE compared with an antegrade wire escalation strategy.

The secondary endpoints are: (1) technical and procedural success4-6; (2) total procedure time (defined as the interval between administration of local anesthesia for obtaining vascular access and removal of the last catheter); (3) fluoroscopy time to cross the CTO and total fluoroscopy time; (4) total air kerma radiation exposure; (5) total contrast volume; and (6) number of wires, microcatheters, balloons, and stents used.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Willing and able to give informed consent
* Undergoing clinically-indicated CTO PCI with a planned antegrade crossing approach

Exclusion Criteria:

* Plan for primary retrograde approach for CTO crossing
* Ostial CTOs (within 5 mm of vessel ostium)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2015-09; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | Until Hospital Discharge (usually 1 day after procedure)
  Incidence of procedural major adverse cardiovascular events (MACE, composite death, emergent coronary artery bypass graft surgery, tamponade requiring pericardiocentesis, and stroke)

SECONDARY OUTCOMES:
Procedure time to Cross the CTO | Until end of procedure (usually 2-3 hours after procedure starts)
Technical and procedural success | Until end of procedure (usually 2-3 hours after procedure starts)
Total procedure time | Until end of procedure (usually 2-3 hours after procedure starts)
  Interval between administration of local anesthesia for obtaining vascular access and removal of the last catheter)
Fluoroscopy time to cross CTO and total fluoroscopy time | Until end of procedure (usually 2-3 hours after procedure starts)
Total air kerma radiation exposure | Until end of procedure (usually 2-3 hours after procedure starts)
Total contrast volume | Until end of procedure (usually 2-3 hours after procedure starts)
Number of wires, microcatheters balloons and stents used. | Until end of procedure (usually 2-3 hours after procedure starts)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil S Brilakis, MD, PhD, Study Chair — North Texas Veterans Healthcare System
Locations (11):
- United States (11):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - United Heart and Vascular Clinic and United Hospital, Saint Paul, Minnesota
  - Missouri Heart Center, Columbia, Missouri
  - St. Luke's Mid America Heart Institute, Kansas City, Missouri
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Wellspan Heart and Vascular, York, Pennsylvania
  - North Central Heart/Avera Heart Hospital, Sioux Falls, South Dakota
  - VA North Texas Healthcare System, Dallas, Texas
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Background] Michael TT, Papayannis AC, Banerjee S, Brilakis ES. Subintimal dissection/reentry strategies in coronary chronic total occlusion interventions. Circ Cardiovasc Interv. 2012 Oct;5(5):729-38. doi: 10.1161/CIRCINTERVENTIONS.112.969808. PMID 23074346
- [Background] Wosik J, Shorrock D, Christopoulos G, Kotsia A, Rangan BV, Roesle M, Maragkoydakis S, Abdullah SM, Banerjee S, Brilakis ES. Systematic Review of the BridgePoint System for Crossing Coronary and Peripheral Chronic Total Occlusions. J Invasive Cardiol. 2015 Jun;27(6):269-76. PMID 26028653